CLINICAL TRIAL: NCT03195660
Title: Adherence to ASV Therapy in Heart Failure With Preserved Ejection Fraction Feasibility Study
Acronym: CAT-PEF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding for study was withdrawn
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-16-12-01
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Results first posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-04

CONDITIONS: Heart Failure With Normal Ejection Fraction; Sleep Apnea
Keywords: adaptive servo-ventilation; ASV; HFpEF
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: Prospective, single-arm, un-blinded, multi-center
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- ASV Therapy (Experimental): ASV Therapy
  Interventions: Device: ASV Therapy

INTERVENTIONS:
Device: ASV Therapy — AirCurve 10 ASV device set up in AutoSet mode
  Other Names: AirCurve 10 ASV

SUMMARY:
This study is designed to demonstrate feasibility of study conduct and that acceptable adherence to adaptive servo-ventilation (ASV) therapy can be achieved in recently hospitalized HFpEF patients with moderate to severe sleep apnea. All subjects meeting the criteria will receive ASV therapy.

DETAILED DESCRIPTION:
Cardiovascular Improvements with Minute Ventilation-targeted ASV Therapy in Heart Failure Study (CAT-HF) was a randomized controlled clinical trial in the United States and Germany. It was designed to evaluate the effect of ASV in hospitalized heart failure (HFrEF and HFpEF) patients on a global rank endpoint of survival free from CV hospitalization and improvement in functional capacity measured by 6-minute walk distance. Analysis of the 126 subjects that were randomized showed a neutral result for the primary endpoint; however, in the pre-specified analysis of the primary endpoint by LVEF strata, there was a favorable statistically significant difference in the HFpEF subgroup (p=0.036).

Although the CAT-HF study showed a positive signal in the HFpEF subgroup, these patients represented a small percentage of the randomized subjects in the study. The current study aims to show that by applying newer technologies to support adherence, as well as focusing on the lessons learned in CAT-HF to identify and recruit HFpEF patients, acceptable adherence to ASV therapy can be achieved in HFpEF patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years or older
2. Patients with heart failure with preserved ejection fraction (HFpEF; LVEF ≥50%)
3. Hospital admission or equivalent (such as ER visit alone or clinic visit alone) and acute decompensated HF as determined by:

   1. Dyspnea at rest or with minimal exertion AND
   2. Treatment with at least one dose of IV diuretic or ultrafiltration AND
   3. At least two of the following signs and symptoms:

   i. Orthopnea ii. Pulmonary rales that do not clear with cough iii. Congestion on chest X-ray iv. Local BNP or NT pro-BNP level: A. No current atrial fibrillation (AFib): BNP≥100 pg/mL or NT pro- BNP≥300 pg/mL OR B. Current AFib: BNP≥150 pg/mL or NT pro-BNP≥450 pg/mL
4. Sleep disordered breathing (SDB) documented by screening polygraphy with an AHI≥15 events/hour (e/hr)
5. Patient is able to fully understand study information and sign informed consent

Exclusion Criteria:

1. Right-sided heart failure without left-sided failure
2. Current chronic use (within 4 weeks of study entry) of any PAP therapy (eg, CPAP, APAP, or bi-level) or contraindicated for PAP therapy
3. Sustained systolic blood pressure <80 mmHg at baseline
4. Complex congenital heart disease
5. Constrictive pericarditis
6. Chronic hypoxemia as evidenced by sustained oxygen saturation ≤ 85% at rest during the day or at start of nocturnal oximetry recording or regular use of oxygen therapy (day or night)
7. Transient ischemic attack (TIA) or Stroke within 3 months prior to study entry
8. Definite clinically evident acute myocardial infarction within 3 months of study entry
9. Known amyloidosis, hypertrophic obstructive cardiomyopathy, or arteriovenous fistulas
10. Moderate or greater valvular heart disease as the primary reason for heart failure
11. Pregnant, or planning to become pregnant during the study period
12. In the opinion of the investigator, the index acute decompensated HF event was due primarily to uncontrolled AFib with fast ventricular response rate
13. Inability to comply with planned study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2017-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher O'Connor, MD, Study Chair — Inova Heart and Vascular Institute
Locations (4):
- United States (3):
  - University of California San Diego, San Diego, California
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Inova Heart and Vascular Institute, Falls Church, Virginia
- Heart and Diabetes Center - West Rhine-Westphalia, Bad Oeynhausen, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Six participants overall were consented for the study, and baseline data on these participants was collected at the baseline visit. Following on from this, four participants did not meet the entry criteria for the study. Two participants started ASV therapy, but the study was terminated before the follow up period.
Period: Overall Study
Arm/Group | ASV Therapy
Started | 2
Completed | 0
Not Completed | 2
Not completed — The study was terminated | 2

BASELINE CHARACTERISTICS:
Population: Six participants overall were consented for the study, and baseline data on these participants was collected at the baseline visit. Following on from this, four participants did not meet the entry criteria for the study. Two participants started ASV therapy, but the study was terminated before the follow up period.
Arm/Group | ASV Therapy
Number analyzed (Participants) | 6
Age, Continuous [Mean (Full Range); unit: years] | 63 [42 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6
Ejection fraction [Mean (Full Range); unit: percent] | 64.5 [55 to 71]

OUTCOME MEASURES:

1. Primary Outcome: ASV Adherence
Description: Average hours used per day
Time Frame: 3 months
Population: The study was terminated prior to the follow-up period
Arm/Group | ASV Therapy
Number analyzed (Participants) | 0

2. Secondary Outcome: KCCQ-12
Description: Change in KCCQ-12 score. Cardiomyopathy Questionnaire (Kansas City) (KCCQ-12) is a short questionnaire to evaluate quality of life in heart failure patients. All scores are scaled from 0-100 where low scares represent very poor health and high scores represent excellent health.
Time Frame: 3 months
Population: The study was terminated prior to the follow-up period
Arm/Group | ASV Therapy
Number analyzed (Participants) | 0

3. Secondary Outcome: Hospitalizations
Description: Number of hospitalizations per subject
Time Frame: 3 months
Population: The study was terminated prior to the follow-up period
Arm/Group | ASV Therapy
Number analyzed (Participants) | 0

4. Secondary Outcome: Death
Description: Number of deaths
Time Frame: 3 months
Population: The study was terminated prior to the follow-up period
Arm/Group | ASV Therapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | ASV Therapy
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
Study was terminated early; results were not analyzed.

Six participants overall were consented for the study; four participants did not meet the entry criteria for the study. Two participants started ASV therapy, but the study was terminated before the follow up period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-28): https://cdn.clinicaltrials.gov/large-docs/60/NCT03195660/Prot_SAP_000.pdf